CLINICAL TRIAL: NCT02984202
Title: Phase I Safety Study for a New Two-Shank Auditory Midbrain Implant (AMI)
Brief Title: Auditory Midbrain Implant Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hannover Medical School (Other)
Collaborators: University of Minnesota (Other); Cochlear (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NIH U01 DC013030
Record Dates: First submitted 2016-11-21; First posted 2016-12-06 (Estimated); Last update posted 2020-08-03 (Actual); Status verified 2020-07

CONDITIONS: Deafness; Perception
MeSH Terms: conditions — Hearing Loss, Sensorineural

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Safety/Efficacy (Experimental): Patients will be implanted with the AMI and evaluated for safety and efficacy over a 2-year period. The placement of the AMI array into the inferior colliculus will also be evaluated.
  Interventions: Device: auditory midbrain implant (AMI)

INTERVENTIONS:
Device: auditory midbrain implant (AMI)

SUMMARY:
The objectives of the clinical study are to implant five deaf patients (those with Neurofibromatosis Type II, NF2) with a new two-shank auditory midbrain implant array (AMI; developed by Cochlear Limited) into the central nucleus of the inferior colliculus in order to assess the safety, reliability, consistency of placement, and performance of the AMI device. The clinical trial is being performed at Hannover Medical School in Germany in collaboration with University of Minnesota (USA) and Cochlear Limited (Australia). The clinical trial is being managed by Hannover Clinical Trial Center in Germany.

DETAILED DESCRIPTION:
Cochlear implants are used in the cochlea (part of the inner ear) where they send electrical signals for activation of the auditory nerve to restore hearing to deaf patients. For patients without a functioning auditory nerve, there is an auditory brainstem implant (ABI), which is placed on the surface of the brainstem in a more central location to restore hearing. Unfortunately, the hearing performance of the ABI is typically lower than the performance of the cochlear implant. There are several reasons for the lower success of the ABI. Due to the tumor and/or tumor removal process for the NF2 condition, there is potential damage caused at the brainstem level that has been linked to the poorer performance. The anatomical changes caused by the tumor also make it difficult to properly visualize and place the ABI surface array into the correct location. In addition, if there is a large tumor that needs to or has been removed, then there can be a large cavity in the brainstem space with the possibility that the ABI surface array can move from its initial location over time.

Therefore, for the past 16 years, a new implant has been developed in an international collaboration that presents electrical stimuli into a midbrain region, the inferior colliculus. This new implant is called the auditory midbrain implant (AMI). The current version consists of two shanks with with 11 electrode contacts linearly spaced along each shank. The two shanks are inserted into the inferior colliculus to align the electrodes along different pitch layers to be able to stimulate them individually with varying temporal pulse patterns.

In the period from 2006 to 2010, a former version of the current AMI was implanted and evaluated in five NF2 deaf patients for hearing restoration. This first AMI implant consisted of only one shank in contrast with the current two-shank array. Encouragingly, the clinical trial at that time showed that the AMI was safe for all five patients. All patients achieved improvements in their hearing capacity, especially in the form of environmental sound awareness and lip-reading enhancement. One patient additionally attained good speech perception that is within the upper range of ABI NF2 patients. However, this speech perception is not yet at the level that can be attained in cochlear implant patients.

Based on these experiences and additional studies in animals, we have developed the second version of the AMI that consists of two shanks that will be implanted into the inferior colliculus and is expected to provide significant improvements in hearing performance compared to the previous AMI by stimulating more effectively across the three-dimensional inferior colliculus.

The purpose of this clinical trial is to evaluate the safety, reliability, and performance of the new two-shank AMI in deaf NF2 patients. The ability to consistency place the AMI array into the inferior colliculus will also be evaluated.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 and ≤75 years
2. Diagnosis of NF2 (i.e., Neurofibromatosis Type 2)
3. Bilateral deafness without a functional auditory nerve or insufficient residual hearing while being ineligible for cochlear implant
4. Eligible for brainstem or midbrain surgery for a standard clinical procedure, including to remove a tumor, replace or reposition an existing ABI, or implant a new ABI
5. No or minimal benefit from a previously implanted auditory brainstem implant (ABI) (i.e. patient has requested an alternative hearing option due to insufficient benefit on a daily basis); or poor performance expected with an ABI due to a high risk of array movement associated with removal of a large tumor or anatomical abnormalities/damage (e.g., associated with altered development, tumor compression, radiation therapy, surgical intervention, or other treatments)
6. No further lesions of the auditory pathway from the inferior colliculus (IC) to the auditory cortex
7. Post-linguistic onset of contralateral severe-to-profound neural hearing loss
8. Women with childbearing potential: willingness to use a reliable contraceptive method (e.g. copper intrauterine devices or hormonal methods) after consulting their gynecologists
9. Written informed consent

Exclusion Criteria:

1. Medical, neurological, or psychological conditions that would contra-indicate undergoing surgery, e.g. acute cardiac infarction, history of stroke, dementia
2. Additional handicaps that would prevent participation in evaluations
3. Pregnant and breast feeding woman, prisoners, or anyone in custody
4. Known allergies to one of the components of the implant
5. Other active devices with potential interference with brain implants, such as transcranial magnetic stimulators
6. Additionally, in the event of other serious diseases (e.g. progressive carcinoma or chronic renal failure) the investigators will decide on a case-by-case basis whether to enroll the patient in the trial

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2016-10-17 (Actual); Primary Completion 2020-06-25 (Actual); Study Completion 2020-06-25 (Actual)

PRIMARY OUTCOMES:
Collection of serious adverse events of AMI | 24 months
  Collection of investigational device related serious adverse events during the evaluation period.
Position of AMI array in midbrain | 24 months
  Evaluation of the final position of the two shanks of the AMI array in the inferior colliculus which includes angles and insertion locations of each shank relative to specific anatomical landmarks. The frequency/pitch ordering of the sites along each shank will also be measured which provides how many electrode sites are correctly positioned into the inferior colliculus and thus the depth location of each shank relative to the surface of the midbrain. All of these measurements provide the final position of the AMI array in the midbrain.

SECONDARY OUTCOMES:
Speech perception performance of AMI | 24 months
  Relative difference of the speech perception score between current ABI recipients with NF2 (collected data from the same clinical site) and AMI recipients with NF2 at the two-year post-operative evaluation visit.

CONTACTS AND LOCATIONS:
Locations (1):
- Hannover Medical School, Hanover, Lower Saxony, Germany